CLINICAL TRIAL: NCT04355026
Title: Use of Bromhexine and Hydroxychloroquine for Treatment of COVID-19 Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General and Teaching Hospital Celje (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBCebromhexinCovid-19
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxychloroquine and bromhexine (Experimental): Bromhexine 16 mg TID + hydroxychloroquine 200 mg BID
  Interventions: Drug: Bromhexine Oral Tablet and/or hydroxychloroquine tablet
- hydroxychloroquine alone (Active Comparator): hydroxychloroquine 200 mg BID
  Interventions: Drug: Bromhexine Oral Tablet and/or hydroxychloroquine tablet

INTERVENTIONS:
Drug: Bromhexine Oral Tablet and/or hydroxychloroquine tablet — bromhexine 16 mg TID hydroxychloroquine 200 mg BID
  Other Names: hydroxychloroquine

SUMMARY:
In the current situation it is of great importance to discover a safe, cost-effective and available treatment strategy in order to limit the rapidly spreading SARS-Cov-2. Recent studies have shown that hydroxychloroquine could have a role in the treatment of infected patients. It is however not very likely that hydroxychloroquine alone could be adequate for treatment of Covid-19 disease. Effective therapy that prevents the virus entrance should contain at least TMPRSS2 inhibitor or a competitive inhibitor of viral ACE 2 binding. The use of bromhexine at the dose adequate to selectively inhibit the TMPRSS2, resulting in preventing of viral entrance via TMPRSS2-specific pathway, coud be an effective treatment of Covid-19. In our study we would like to explore the therapeutic potential of bromhexin and hydroxychloroquine in Covid-19 patients.

Hypothesis

1. Combined treatment with bromhexin and hydroxychloroquine shortens the course of disease in hospitalized Covid-19 patients compared to hydroxychloroquine alone.
2. Combined treatment with bromhexin and hydroxychloroquine lowers the incidence of secundary pulmonary infections in hospitalized Covid-19 patients compared to hydroxychloroquine alone.
3. Combined treatment with bromhexin and hydroxychloroquine decreases the need for ICU admission in hospitalized Covid-19 patients compared to hydroxychloroquine alone.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* confirmed infection (positive PCR from nasopharyngeal swab),
* fullfilled hospital admission criteria

Exclusion Criteria:

* pregnancy,
* known allergy for bromhexine or hydroxychloroquine,
* epilepsy,
* prolonged QTc interval,
* Child C liver disease,
* dementia,
* psychoorganic syndrome,
* terminal chronic disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization | through study completion, an average of 6 months
  number of days the patient is treated in the hospital
Duration of disease | through study completion, an average of 6 months
  Number of days from the onset of symptoms to hospital discharge

SECONDARY OUTCOMES:
Hospital-aquired pneumonia | through study completion, an average of 6 months
  Incidence of HAP
ICU stay duration | through study completion, an average of 6 months
  Number of days spent in the ICU
Oxygene therapy duration | through study completion, an average of 6 months
  number of days on oxygene therapy
Mechanical ventilatory support duration | through study completion, an average of 6 months
  Number of hours on mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- SB Celje, Celje, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided